CLINICAL TRIAL: NCT07096531
Title: The Effectiveness of Suit Therapy With Dual Task Exercises on Gross Motor Functions and Walking in Children With Diplegic Cerebral Palsy
Brief Title: Effectiveness of Suit Therapy With Dual Task Exercises on Gross Motor Functions and Walking in Children With Diplegic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Waleed Saleh Althobaiti, B.Sc. in Physical Therapy, Faculty of Physical Therapy, Kafrelsheikh University, Kafrelsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-533
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Suit Therapy; Dual Task Exercises; Gross Motor Functions; Walking; Children; Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Active Comparator): Patients will receive suit therapy.
  Interventions: Other: Suit therapy
- Group (B) (Experimental): Patients will receive suit therapy in addition to dual-task exercises.
  Interventions: Other: Suit therapy + Dual-task exercises

INTERVENTIONS:
Other: Suit therapy — Patients will receive suit therapy.
  Arms: Group (A)
Other: Suit therapy + Dual-task exercises — Patients will receive suit therapy in addition to dual-task exercises.
  Arms: Group (B)

SUMMARY:
This study aims to investigate the effect of suit therapy combined with dual-task training on gross motor performance and walking abilities in children with diplegic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a non-progressive motor impairment syndrome caused by brain defects or lesions that occur in an immature brain before, during, or within two years after birth.

Therapeutic approaches for CP include neurodevelopmental treatment, Vojta therapy, sensory integration therapy, and conductive education. Specific therapeutic strategies for CP may differ, but they all aim to improve the independence of children with CP.

Suit therapy is a relatively new and experimental form of therapy designed to help those with cerebral palsy improve muscle tone, posture, and movements.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 12 years.
* Both sexes.
* A medical diagnosis of spastic diplegic CP made by pediatricians or pediatric neurologists.
* Children with spasticity grades ranged from 1 to 2+ according to the Modified Ashworth scale (MAS).
* Children who can sit on the chair with good balance and recognize and follow verbal orders and commands are included in both testing and training techniques.

Exclusion Criteria:

* They had a permanent deformity (bony or soft tissue contractures).
* Children having visual or auditory defects.
* Current hospitalization for urgent medical reasons.
* Severe mental retardation.
* Children who will undergo fewer than twelve regular sessions of physical therapy at their place will not be included in the survey.
* Children with a history of epileptic seizure or any diagnosed cardiac or orthopedic disability that may hinder assessment methods and treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Gross Motor Function Measure 88 (GMFM-88) | 3 months post-exercise
  The Gross Motor Function Measure (GMFM) 88 will be used to determine the severity of each case and to assess the child's motor performance in five dimensions: lying and rolling (17 items); sitting (20 items); crawling and kneeling (14 items); standing (13 items); and walking, running, and jumping (24 items). All items will be checked and scored before interpretation of the child's performance in each dimension. Scores of each dimension will be expressed as a percentage of the maximum scores for that dimension. The total score will be obtained by averaging the percentage scores across the five dimensions. Individual dimensions of GMFM-88 can be administered depending on the child's current level of function.

SECONDARY OUTCOMES:
Evaluation of balance using the Pediatric Balance Scale (PBS) | 3 months post-exercise
  The Pediatric Balance Scale (PBS) is a standardized tool for testing balance. The items can be measured within 15 minutes and do not require specialized equipment. The Pediatric Balance Scale is a modified version of the Berg Balance Scale, used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function), with a maximum score of 56 points

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.